CLINICAL TRIAL: NCT01703715
Title: Hydration and Outcome in Older Patients
Acronym: HOOP
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 12029
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Dehydration
Keywords: Hydration; Elderly patients; Age 65 years and over; Admitted acutely to medical admissions ward
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants provide 5mls of whole blood on admission, at 48 hours post admission and at 3 month following discharge. This blood is to be analysed for urea, creatinine, sodium, potassium, osmolality, full blood count as well as renin and aldosterone.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients aged 65 years and over: All patients aged 65 years and over admitted to acutely to medical wards
  Interventions: Device: The Hydrant

INTERVENTIONS:
Device: The Hydrant — The Hydrant is a new form of "drinking system" that may be used to provide continuous access to hydration will be given to 20 patients. 10 of the patients will have mild cognitive impairment with Mini Mental State Examination less than 24 and 10 with normal cognitive function. Patients and staff will be interviewed to assess the feasibility of the hydrant.

SUMMARY:
Dehydration is recognised as a major issue in healthcare. Recovery after illness, extended length of stay, pressure sores and slow tissue recovery can all be impacted by dehydration. One of the biggest problems for many people with regard to getting a drink is easy, independent access - if they can't reach the jug/cup without a struggle then they often will go thirsty and potentially become dehydrated.

The purpose of this study is to investigate the impact of dehydration on outcome in patients 65 years and over. Furthermore we aim to assess the impact of providing easy, 24 hour, independently accessible fluids on reducing dehydration as well as improving patient experience.

We hypothesise that patients who are dehydration will take longer to recover from illness and stay in hospital for longer periods.

ELIGIBILITY:
Inclusion Criteria:

1. - All patients of 65 years and over that are admitted acutely to medical wards
2. - Ward staff who have been working in the clinical area for the duration of the trial (The Hydrant part of the study).

Exclusion Criteria:

1. - Patients who are moribund
2. - Patients who are doubly incontinent
3. - Patients on the end of life pathway
4. - Patients with terminal illness with a known life expectancy less than 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients admitted acutely to medical wards who are aged 65 years and over.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Serum Osmolality | At admission and 48hrs post admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N Lobo, MD, FRCS, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom